CLINICAL TRIAL: NCT05532865
Title: Prospective Cohort of Patients With Systemic Sclerosis at Brest University Hospital and Constitution of a Biobank
Brief Title: Prospective Cohort of Patients With Systemic Sclerosis at Brest University Hospital With Biobanking
Acronym: SCLEROBREST
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC21.0258
Record Dates: First submitted 2022-09-05; First posted 2022-09-08 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Systemic Sclerosis
Keywords: Systemic Sclerosis; Patient library
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood samples 80 ml of blood samples collected at inclusion and at 18 months ((60 ml for Peripheral blood mononuclear cell, 6 ml for plasma, 6 ml for sero, 6 ml for DNA and 2.5 ml for RNA)
  Stool samples A stool sample for collection of digestive microbiota at inclusion
  Skin swab samples A skin swab sample for collection of skin microbiota at inclusion and at 18 months
  Skin biopsy (optional) at inclusion and at 18 months
  Questionnaires on quality of life, pain and disability At inclusion and each year for 5 years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with systemic sclerosis: It is a descriptive cohort of systemic sclerosis patients
  Interventions: Other: Blood samples; Other: Stool samples; Other: Skin swab samples; Other: Questionnaires on quality of life, pain and disability; Other: Skin biopsies

INTERVENTIONS:
Other: Blood samples — 80 ml of blood samples collected at inclusion and at 18 months
Other: Stool samples — A stool sample for collection of digestive microbiota at inclusion
Other: Skin swab samples — A skin swab sample for collection of skin microbiota at inclusion and at 18 months
Other: Questionnaires on quality of life, pain and disability — At inclusion and each year for 5 years
Other: Skin biopsies — At inclusion and 18 months

SUMMARY:
This study corresponds to a monocentric prospective cohort of adult patients with systemic sclerosis.

It will allow the constitution of an organized collection of longitudinal clinical data as well as collection of biological samples, including blood samples, as well as stool sample and skin swab for microbiota analysis.

ELIGIBILITY:
Inclusion Criteria:

* Major patient with systemic sclerosis defined according to the EULAR 2013 criteria (see Appendix 1)
* Patient evaluated within the framework of the reference center for rare autoimmune diseases of the CHU of Brest.
* Patient affiliated to the social security system
* Patient having signed a written informed consent.

Exclusion Criteria:

* Minor
* Patient under legal protection (guardianship, curatorship)
* Refusal to participate
* Patient unable to consent
* Pregnant or breastfeeding woman
* Hemoglobin (Hb) level < 7g/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major patient with systemic sclerosis defined according to the EULAR 2013 criteria
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2032-10-13 (Estimated); Study Completion 2032-10-13 (Estimated)

PRIMARY OUTCOMES:
Age | 5 years
  To assess whether age correlates with disease profile and progression
Sex | 5 years
  To assess whether sex correlates with disease profile and progression
Weight | 5 years
  To assess whether weight correlates with disease profile and progression
Medical history | 5 years
  To assess whether medical history predicts the pattern and course of the disease
Family history | 5 years
  To assess whether family history predicts the pattern and course of the disease
Rodnan score | 5 years
  This score evaluates the thickness of the skin from 0 to 51. 0 meaning the absence of scleroderma (the healthiest score) and 51 completely sclerotic skin (the worst possible score)
active digital ulcers | 5 years
  4 characteristics must be taken into account:
  1. the type of ulcer: mechanical/on calcinosis/ischemic
  2. the recent/semi-recent/chronic character,
  3. the painful character or not,
  4. the total number of fingers affected on the 10 fingers.
dyspnea | 5 years
  * stage I: absence of dyspnea for usual efforts: no discomfort is felt in everyday life,
  * stage II: dyspnoea for usual heavy exertion, such as brisk or hill walking or climbing stairs (≥ 2 floors),
  * stage III: dyspnea for low intensity efforts of everyday life, such as walking on flat ground or climbing stairs (< 2 floors),
  * stage IV: permanent dyspnea at rest or for minimal effort (putting on a garment, for example)
Free Carbon Monoxide Diffusion (DLCO) | 5 years
  Free Carbon Monoxide Diffusion (DLCO) in percentage.
6-minute walk test | 5 years
  Distance (in meters) covered in the 6-minute walk test.
systemic pulmonary arterial pressures | 5 years
  Measured on cardiac ultrasound.

SECONDARY OUTCOMES:
SF-36 (Short-Form 36) | 5 years
  The SF-36 is an indicator of health status and quality of life. The SF-36 has eight dimensions; the scores are weighted sums of the questions in each section. This scores range from 0 - 100. Lower scores indicate more disability and higher scores less disability.
  The eight dimensions of this score are:
  * Vitality
  * Physical functioning
  * Bodily pain
  * General health perceptions
  * Physical role functioning
  * Emotional role functioning
  * Social role functioning
  * Mental health
BPI : Pain scale | 5 years
  A quick and easy way to measure the intensity of pain and its impact on daily activities. Patients rate the maximum, minimum, average and current intensity of their pain and the influence of pain on seven aspects of functional ability. 3 scores are obtained between 0 and 10, with 10 corresponding to :
  * the worst pain experienced in the last 24 hours
  * the highest pain intensity combining the most intense, the least intense, the average pain and the pain experienced at the time of the questionnaire
  * the highest interference of the pain on daily activities
HAQ- Health Assessment Questionnaire - Disability Index | 5 years
  Evolution of HAQ-DI (Health Assessment Questionnaire - Disability Index) during follow-up 8 fields questionnaire (DRESSING & GROOMING, ARISING, EATING, WALKING, HYGIENE, REACH, GRIP, Other activities), scaled from 0 to 3, 3 meaning a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement